CLINICAL TRIAL: NCT03513809
Title: Spontaneous Breathing and Progression of Lung Injury in Acute Respiratory Distress Syndrome Before Connection to Mechanical Ventilation
Brief Title: Inflammation and Distribution of Pulmonary Ventilation Before and After Tracheal Intubation in ARDS Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Pontificia Universidad Catolica de Chile (Other)
Collaborators: Comisión Nacional de Investigación Científica y Tecnológica (Other Government)
Responsible Party: Principal Investigator, Jaime Retamal, Medical Doctor, Pontificia Universidad Catolica de Chile
Other Study IDs: 170315007; 1171810 (Other Grant/Funding Number: FONDECYT)
Record Dates: First submitted 2018-04-19; First posted 2018-05-02 (Actual); Last update posted 2021-03-10 (Actual); Status verified 2021-03

CONDITIONS: Acute Hypoxemic Respiratory Failure; Acute Respiratory Distress Syndrome
Keywords: Acute Hypoxemic Respiratory Failure; Acute Respiratory Distress Syndrome; Electrical impedance tomography; Spontaneous breathing; Ventilation induced-lung injury; Patient self-inflicted lung injury
MeSH Terms: conditions — Respiratory Insufficiency; Respiratory Distress Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Days
Biospecimen Retention: Samples Without DNA — Plasma samples and bronchoalveolar lavage samples.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Acute hypoxemic respiratory failure: Patients with acute hypoxemic respiratory failure breathing spontaneously with no requirements of immediate intubation connected to thoracic electrical impedance tomography.
  Interventions: Device: Thoracic electrical impedance tomography

INTERVENTIONS:
Device: Thoracic electrical impedance tomography — Non invasive, radiation-free, bedside monitoring tool for distribution of pulmonary ventilation.

SUMMARY:
Spontaneous breathing efforts in patients with respiratory failure connected to mechanical ventilation, has been associated with strong respiratory muscles activity. However, these mechanisms may will be present in patients with acute lung deseases who are breathing with no ventilatory support.

We hypothesize that spontaneous breathing during acute respiratory failure could induced lung inflammation and worsen lung damage. Hereby, the connection to a ventilatory support tool, may protect the lungs from spontaneous ventilation-induced lung injury.

To test our hypothesis, our aim is to determine the effects of spontaneous breathing in acute respiratory failure patients, on lung injury distribution; and to determine whether early controlled mechanical ventilation can avoid these deleterious effects by improving air distribution.

DETAILED DESCRIPTION:
Prospective clinical protocol in patients admitted to the ICU of the Hospital Clínico UC-Christus, Santiago de Chile, with diagnosis of acute hypoxemic respiratory failure, but who are still ventilating spontaneously.

Clinical data:

After hospital admission, patients who meet inclusion/exclusion criteria will be asked to consent to participate in the study protocol. Patients will be monitored conventionally according with hospital protocols (continuous ECG, SpO2, invasive arterial pressure, and intermittent arterial blood gases).

EIT Monitoring:

An EIT belt will be installed around the patient thorax connected to Enlight impedance tomography monitor (Dixtal, São Paulo, Brazil). EIT data will be recorded during periods of 3 minutes for offline analysis. Regional distribution of ventilation will be analyzed by dividing the image in four ROIs, each covering 25% of the ventro-dorsal distance encompassing the whole lung area. In addition we will estimate recruitment-derecruitment, and overdistention, regionally. In addition, pendelluft phenomena, and spatial patterns of regional deformation will be assessed.

Study protocol:

After patient inclusion, the first EIT and physiological data acquisition will be recorded (hemodynamics, respiratory variables, arterial blood gases, plasma samples). The data acquisition will be repeated every 6 hours from enrollment until intubation, or upto 24 hours of follow up, after which the patient will only be followed for clinically relevant outcomes. If within 24 hours of inclusion the attending physician decides intubation and connection to MV, an extra assessment of EIT, clinical data and blood samples will be performed. After intubation these assessments will include MV data and will be repeated hourly for the first 6 hours, and then at 12, 18 and 24 hours thereafter.

Bronchoalveolar lavages:

Immediately after intubation and initial stabilization, a fiberoptic bronchoscope-guided distal-protected small volume bronchoalveolar lavage (FODP mini-BAL) will be performed. This early BAL will be used as representative of the previous period of spontaneous ventilation. After 48 hours of controlled MV a new BAL will be performed, at the same regions than the first BAL, to compare the changes in the pattern of regional inflammation. For each BAL one or two aliquots of 20 ml of warmed (37°C) sterile isotonic saline will be administered and subsequently recovered in dorsal (lateral inferior) and ventral segments (medial lobe or lingula). The first recovered aliquot will be discarded while the remaining BAL fluid will be rapidly filtered through a sterile gauze and spun at 4°C at 400 x g for 15 min. The supernatant will be centrifuged at 80,000 x g for 30 min at 4°C in order to remove the surfactant-rich fraction and then divided into aliquots and frozen at - 80 °C for subsequent cytokine and mechanotransduction markers determinations.

* BAL samples will only be collected if the attending physician determines that this procedure is clinically necessary.

Cytokine analysis in serum, BALF and tissue supernatants:

Quantification of TNF-α, IL-1β, IL-6, IL-8 and IL-10 levels in plasma at time to inclusion, intubation, and 24 and 48 hours after intubation. BALF will be analyzed to determine quantification of neutrophils, cytokines (TNF-α, IL-1β, IL-6, IL-8 and IL-10) and TGF-β (extracellular cytokine with mechanotransduction proprieties) at intubation time and 48 hours after intubation.

Gas Exchange, Hemodynamics, and Ventilatory Data:

At each time of physiological acquisition we will collect arterial and central venous blood gases (if central venous catheter is present). We will assess hemodynamics (arterial blood pressure, central venous pressure, central venous pressure inspiratory swings, heart rate), and ventilatory parameters. While patients remain in spontaneous ventilation we will assess respiratory rate, ventilatory pattern, and Borg dyspnea score. After intubation and connection to MV we will collect full ventilatory data from the pneumotach system for later analysis of flows, pressures and volumes.

Statistical Analysis:

For the clinical protocol we don´t have previous data about distribution of ventilation between dependent and non-dependent lung regions during spontaneous ventilation. Therefore, we calculated sample size based on an expected effect size of 0.5, with a standard deviation two times larger, between the period of spontaneous ventilation before intubation, and the period of controlled MV after intubation. For a power of 0.8 and a two-sided error of 0.05 the calculated sample size is 32. However, of the included patients, only a fraction will be intubated, so we calculated that 60 to 80 patients must be included during the 4-year period, to complete the required number of patients available for before-after analysis. We will express values as means - standard deviation (SD) or median - range where appropriate. The Shapiro-Wilk test will be used to test data for normality. Groups will be compared using Student's t-test or Mann-Whitney U-test, one-way (repeated-measures) analysis of variance (ANOVA) or Kruskal- Wallis test. Interactions between groups and time will be assessed with two-way repeated-measures ANOVA. The Bonferroni adjustment for multiple tests will be applied for post hoc comparisons. The statistical analyses will be conducted by SPSS v.20.0.0 software (SPSS, Inc, Chicago, IL, USA), and GraphPad Prism version 5.0 (GraphPad Software, San Diego, CA, USA).

ELIGIBILITY:
Inclusion Criteria:

* Acute respiratory symptoms for less than seven days
* Acute hypoxemic respiratory failure defined by a ratio of partial pressure of arterial oxygen (Pao2) to Fio2 of 300 mm Hg or less, while breathing with standard oxygen mask at FiO2 > or equal to 30%
* Increased work of breathing defined by either:

  i. Respiratory rate > 25 / min, or ii. Signs of intercostal or supraclavicular retraction
* Less than 24 hours since criteria 2 and 3 are met.

Exclusion Criteria:

* Acute respiratory failure secondary to exacerbation of chronic respiratory disease or to cardiogenic pulmonary edema, PaCO2 > 45 mm Hg, decreased conscious level (Glasgow Coma Scale < 13), urgent need for endotracheal intubation, a decision not to resuscitate, and consent refusal.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to the ICU of the Hospital Clínico UC-Christus, Santiago de Chile, with diagnosis of acute hypoxemic respiratory failure, but who are still ventilating spontaneously.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2017-06-08 (Actual); Primary Completion 2021-03-21 (Estimated); Study Completion 2021-03-31 (Estimated)

PRIMARY OUTCOMES:
Inflammation | Plasma: At the time of enrollment and 48 hours post intubation. BALF: Immediately post intubation and 48-96 hours post intubation (only if it is required and indicated by the attending physician).
  Cytokine analysis (TNF-α, IL-1β, IL-6, IL-8 and IL-10) in serum, bronchoalveolar lavage fluid (BALF) and tissue supernatants.

SECONDARY OUTCOMES:
Pulmonary ventilation distribution | Every 6 hours from enrollment to intubation and after connection to mechanical ventilation each hour for the first 6 hours and then at 12, 18, 24 and 48 hours.
  Regional pulmonary ventilation distribution at bedside with electrical impedance tomography

CONTACTS AND LOCATIONS:
Overall Officials: Jaime A Retamal, Principal Investigator — Pontificia Universidad Catolica de Chile
Locations (1):
- Hospital Clínico Universidad Católica, Santiago, Chile

IPD SHARING:
Plan to Share IPD: No
There isn't plan for IPD

REFERENCES:
- [Result] Brochard L. Ventilation-induced lung injury exists in spontaneously breathing patients with acute respiratory failure: Yes. Intensive Care Med. 2017 Feb;43(2):250-252. doi: 10.1007/s00134-016-4645-4. Epub 2017 Jan 10. No abstract available. PMID 28074228
- [Result] Mascheroni D, Kolobow T, Fumagalli R, Moretti MP, Chen V, Buckhold D. Acute respiratory failure following pharmacologically induced hyperventilation: an experimental animal study. Intensive Care Med. 1988;15(1):8-14. doi: 10.1007/BF00255628. PMID 3230208
- [Result] Yoshida T, Uchiyama A, Fujino Y. The role of spontaneous effort during mechanical ventilation: normal lung versus injured lung. J Intensive Care. 2015 Jun 17;3:18. doi: 10.1186/s40560-015-0083-6. eCollection 2015. PMID 27408729
- [Result] Yoshida T, Fujino Y, Amato MB, Kavanagh BP. Fifty Years of Research in ARDS. Spontaneous Breathing during Mechanical Ventilation. Risks, Mechanisms, and Management. Am J Respir Crit Care Med. 2017 Apr 15;195(8):985-992. doi: 10.1164/rccm.201604-0748CP. PMID 27786562